CLINICAL TRIAL: NCT00630773
Title: Feasibility of CPR Adjuncts in Children: Q-CPR Compression Sensor Size Qualification
Brief Title: Q-CPR Compression Sensor Size Qualification in Children
Acronym: PUCK
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Laerdal Medical (Industry)
Responsible Party: Aaron Donoghue, MD, Children's Hospital of Philadelphia
Other Study IDs: 2006-12-5077
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Last update posted 2008-12-03 (Estimated); Status verified 2008-12

CONDITIONS: CPR
Keywords: CPR; compression sensor; chest compression adjuncts

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This prospective, pilot observational study will be performed in the Emergency Department (ED), Pediatric Intensive Care Unit (PICU), Operating Room (OR) and regular inpatient care area (RIPCA) settings at the Children's Hospital of Philadelphia. The differences in trained pediatric health care provider placement of the compression sensor and their assessment of the suitability / willingness to use the current or size modified sensor will be assessed.

DETAILED DESCRIPTION:
Context: Expert recommendations for CPR skills (blowing air into the lungs, pressing on the chest) are poorly followed by health care providers. CPR sensors as small as a hockey "puck" placed on the chest during CPR delivery are able to coach a rescuer to perform better CPR through corrective voice feedback. More adults survive when the quality of CPR (Q-CPR) is improved. This new technology is currently not approved for use in children, specifically 6 months to < 8 years of age.

Objectives:

1. Characterize trained pediatric health care provider opinion concerning how appropriate the current Q-CPR sensor ("puck"), FDA approved for children ≥ 8 years of age, is for use in younger children ages 6m to < 8 years of age.
2. Determine the need for Q-CPR sensor ("puck") size changes to improve its suitability for younger children < 8 years of age, based upon trained pediatric health care provider opinion.
3. Characterize the amount of Q-CPR sensor ("puck") overlap with standard large and small mock defibrillator electrode pads placed in usual locations on the chest.
4. Evaluate trained pediatric health care provider self-reported willingness to use current or modified Q-CPR sensors ("pucks") in younger children, 6 months to < 8 years of age.

Study Design/Setting/Participants: This observational study will be performed in the Emergency Department (ED), Pediatric Intensive Care Unit (PICU), Operating Room (OR) and regular inpatient care area (RIPCA) settings at the Children's Hospital of Philadelphia. Parents and guardians of children ages 6m to < 8 years of age receiving routine clinical care in these patient care areas will be approached for inclusion. Health care practitioners (HCPs) in the ED, OR and PICU will also be approached for inclusion.

Study Measures: Children will have their age, length, weight, and simple measurements of their chest, neck and abdomen taken. The differences in trained pediatric health care provider placement of the compression sensor and their assessment of the suitability / willingness to use the current or size modified sensor will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria - child subjects

  1. Children aged 6 months to 8 years receiving care in the ED, OR, PICU, or RIPCA
  2. Parental or guardian permission (verbal consent), and if appropriate, child assent.
* Inclusion Criteria - HCPs

  1. Physician, nurse, therapist, or technician involved in patient care in the hospital area (ED, OR, PICU, RIPCA) where a consented child subject is located
  2. Verbal consent obtained

Exclusion Criteria:

* child subjects

  1. Obvious chest deformity (pectus excavatum, pectus carinatum) that would make chest dimension measurements difficult or inaccurate.
  2. Absence of child assent as evidenced by either vocal or physical objection to performing measurements.
* HCPs 1. Previous enrollment in the study for a child subject in the same age strata as the subject enrolled at that time

Ages: 6 Months to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Emergency Department (ED), Pediatric Intensive Care Unit (PICU), Operating Room (OR) and Regular Inpatient Care Area (RIPCA) settings at the Children's Hospital of Philadelphia.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2007-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Determination of how appropriate the existing compression sensor is on children aged 6m to 8yrs, based upon trained pediatric health care provider opinion. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Donoghue, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States